CLINICAL TRIAL: NCT00702585
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Comparative Trial to Investigate the Optimal Dose of a Single Administration of Org 36286 (Corifollitropin Alfa) to Induce Monofollicular Ovulation in Women With WHO Group II Anovulatory Infertility
Brief Title: Study to Investigate the Optimal Dose of Org 36286 to Induce Monofollicular Ovulation in Women With WHO Group II Anovulatory Infertility (P07016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07016; 38805
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Infertility
Keywords: Ovulation Induction; Pharmacological effects of drugs; Hormones; Hormone substitutes and Hormone Antagonists; Pharmacological Actions; Randomized; Multi-center; Multi-national
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Org 36286 7.5 µg (Experimental): Org 36286 7.5 µg administered as a single subcutaneous injection on the day of the onset of a spontaneous or progestagen induced withdrawal bleeding or one to two days later.
  Interventions: Drug: Org 36286
- Org 36286 15 µg (Experimental): Org 36286 15 µg administered as a single subcutaneous injection on the day of the onset of a spontaneous or progestagen induced withdrawal bleeding or one to two days later.
  Interventions: Drug: Org 36286
- Org 36286 30 µg (Experimental): Org 36286 30 µg administered as a single subcutaneous injection on the day of the onset of a spontaneous or progestagen induced withdrawal bleeding or one to two days later.
  Interventions: Drug: Org 36286
- Org 36286 60 µg (Experimental): Org 36286 60 µg administered as a single subcutaneous injection on the day of the onset of a spontaneous or progestagen induced withdrawal bleeding or one to two days later.
  Interventions: Drug: Org 36286
- Placebo (Placebo Comparator): Placebo to Org 36286 administered as a single subcutaneous injection on the day of the onset of a spontaneous or progestagen induced withdrawal bleeding or one to two days later.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Org 36286 — Org 36286 single-dose subcutaneous injection
  Other Names: Corifollitropin alpha
  Arms: Org 36286 15 µg; Org 36286 30 µg; Org 36286 60 µg; Org 36286 7.5 µg
Drug: Placebo — Placebo to Org 36286 as a single-dose subcutaneous injection
  Arms: Placebo

SUMMARY:
The objectives of this trial were to investigate the feasibility and the optimal dose of a single administration of Org 36286 to induce monofollicular ovulation in women with WHO Group II anovulatory infertility and to assess the safety (including the absence of antibody formation) of Org 36286.

DETAILED DESCRIPTION:
This was a phase II, randomized, double-blind, placebo controlled, comparative trial to investigate the optimal dose of a single administration of Org 36286 to induce monofollicular ovulation in women with WHO Group II anovulatory infertility.

Treatment injection was given on Day 1-3 after the onset of a spontaneous or progestagen induced withdrawal bleeding. After injection, ultrasound monitoring and sampling for serum hormones were done on treatment Days 3, 5, and daily from Day 7 to 21 or until a urinary luteinizing hormone (LH) peak was detected. From treatment Day 7 the urinary LH response was assessed to detect the preovulatory LH peak. In case of hyperstimulation, production of endogenous gonadotropins could be suppressed by giving daily injections of GnRH antagonist.

Post-treatment assessments were done in the third week after the urinary LH peak. If no LH peak was detected, posttreatment assessments were performed four to five weeks after Org 36286 or placebo injection.

ELIGIBILITY:
Inclusion Criteria:

* Wish to conceive;
* Oligomenorrhea (cycle length >=41 days) or amenorrhea (no menstrual cycle for >6 months);
* Body Mass Index (BMI) >=18 and <=32 kg/m^2;
* Serum FSH levels within normal limits (1-10 IU/L);
* Normal serum prolactin and thyroid stimulating hormone (TSH) levels;
* Progestagen induced withdrawal bleeding or spontaneous menstrual bleeding;

Exclusion Criteria:

* Tumours of the ovary, breast, uterus, pituitary or hypothalamus;
* Pregnancy or lactation;
* Undiagnosed vaginal bleeding;
* Ovarian cysts or enlarged ovaries not related to polycystic ovarian disease (PCOD);
* Any ovarian and/or abdominal abnormality interfering with ultrasound examination;
* Malformations of the sexual organs incompatible with pregnancy;
* Clomiphene resistance with documented anovulation (treated with 150 mg clomiphene for five days and no ovulation);
* Treatment with metformin, gonadotropins, or GnRH analogs within 90 days prior to the start of Org 36286 treatment;
* Treatment with clomiphene citrate within 42 days prior to the start of Org 36286 treatment;
* Alcohol or drug abuse within the 12 months preceding signing of informed consent;
* Any clinically relevant abnormal laboratory value;
* Hypersensitivity to any of the substances in Org 36286;
* Hypersensitivity to Orgalutran® or any of its components;
* Use of any investigational drugs during 90 days before screening or previous participation in this trial.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2001-08-01 (Actual); Primary Completion 2002-10-15 (Actual); Study Completion 2002-10-15 (Actual)

PRIMARY OUTCOMES:
Participant Ovulation Rate in Monofollicular Cycles | Up to 2 Weeks Following LH Peak

SECONDARY OUTCOMES:
Participant Overall Ovulation Rate | Up to 2 Weeks Following LH Pek
Number of Participants With Cancellation of Menstrual Cycle | Up to Day 21
Participant Follicle Size | Up to Day 21
Number of Participants With Miscarriages, Biochemical, Ectopic, Clinical, Vital, Single, or Multiple Ongoing Pregnancies | Up to 10 Weeks Following Ovulation
Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 10 Weeks Following Ovulation
Number of Participants With Clinically Significant Laboratory Abnormalities | Up to 3 Weeks Following Ovulation
Number of Participants With Clinically Significant Changes in Vital Signs | Up to 3 Weeks Followiing Ovulation
Number of Participants With Antibodies to Org 36286 | Up to 3 Weeks Following Ovulation
Participant Serum Follicle Stimulating Hormone (FSH) Level | Up to Day 21
Participant Serum LH Level | Up to Day 21
Participant Inhibin-B, E2, and P Serum Concentration | Up to Day 21
Number of Participants with Ovarian Hyperstimulation Syndrome (OHSS) | Up to 2 Weeks Following LH Peak

REFERENCES:
- [Result] Balen AH, Mulders AG, Fauser BC, Schoot BC, Renier MA, Devroey P, Struijs MJ, Mannaerts BM. Pharmacodynamics of a single low dose of long-acting recombinant follicle-stimulating hormone (FSH-carboxy terminal peptide, corifollitropin alfa) in women with World Health Organization group II anovulatory infertility. J Clin Endocrinol Metab. 2004 Dec;89(12):6297-304. doi: 10.1210/jc.2004-0668. PMID 15579793